CLINICAL TRIAL: NCT00028418
Title: Phase I Study of CL-F-ARA-A in Solid and Hematologic Malignancies
Brief Title: Clofarabine in Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-1972-01; DM93-036; FD-R-001972-01
Record Dates: First submitted 2002-01-04; First posted 2002-01-09 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-11

CONDITIONS: Hematologic Neoplasms; Lymphoproliferative Disorders; Leukemia; Leukemia, Lymphocytic, Chronic
Keywords: Acute Leukemia; Chronic Lymphocytic Leukemia; Antineoplastic Agents; Nucleosides; Dose-Response Relationship, Drug; Cladribine; Fludarabine
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoproliferative Disorders; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Clofarabine

INTERVENTIONS:
Drug: Clofarabine

SUMMARY:
This is a dose-escalation study to determine the maximum tolerated dose and toxic effects of clofarabine in patients with chronic lymphocytic leukemia and other acute leukemias. Clofarabine is a synthesized hybrid nucleoside analog, which is believed to possess the better qualities of fludarabine and chlorodeoxyadenosine, the 2 most active agents against lymphoproliferative disorders. Thus, it is hoped that this drug will be more active and less toxic than similar drugs.

DETAILED DESCRIPTION:
The first group of patients will be treated at the starting dose level of 2 mg/m2 over 1 hour daily for 5 days. Dosage escalation will be permitted in individual patients if no toxicity occurred during the preceding course. Subsequent dose escalations will be by 50% until Grade 2 toxicity, then by 35% until the maximum tolerated dose.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of chronic lymphocytic leukemia
* Diagnosis of other acute leukemia
* At least 2 weeks since prior chemotherapy, immunotherapy, and/or radiotherapy
* Recovered from toxic effects of prior therapy
* Bilirubin no greater than 2 mg/dL
* Creatinine no greater than 1.5 mg/dL

Exclusion criteria:

* Candidate for treatment of higher efficacy or priority
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-02; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M. Kantarjian, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States